CLINICAL TRIAL: NCT01169987
Title: Evaluation of Humira Retention Rate in Psoriasis Patients in Daily Practice and Assessment of Work Productivity and Quality of Life
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-129
Record Dates: First submitted 2010-07-13; First posted 2010-07-27 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Psoriasis
Keywords: Multicenter study
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Treated with Adalimumab: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment is initiated. All medications will be prescribed in the usual manner in accordance with the terms of the marketing authorization and in line with the Belgian reimbursement criteria.

SUMMARY:
This observational study will document to what extent in daily clinical practice Humira (adalimumab) therapy is continued, interrupted or permanently discontinued during a follow-up period of 2 years. Reasons for interrupting or permanently discontinuing Humira therapy and reasons for restarting Humira therapy will be noted. An evaluation will be performed of the effect of the disease on quality of life and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 18 years
* Patient with chronic plaque psoriasis
* Patient newly initiated on Humira
* Patient compliant with Humira Summary of Product Characteristics
* Patient compliant with Belgian reimbursement criteria of Humira in plaque psoriasis
* Patient has signed informed consent

Exclusion Criteria:

* Patients having any of the contraindications mentioned in the Summary of Product Characteristics Humira
* Patients not willing to sign informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis followed in university or peripheral hospitals or peripheral private practices with experience in psoriasis patient care.
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2010-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simonne Lens, MD, Study Director — AbbVie sa

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Treated With Adalimumab: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated. All medications were prescribed in the usual manner in accordance with the terms of the marketing authorization and in line with the Belgian reimbursement criteria.
Period: Overall Study
Arm/Group | Participants Treated With Adalimumab
Started | 191
Completed | 160
Not Completed | 31
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 24
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 133

OUTCOME MEASURES:

1. Primary Outcome: Adalimumab Treatment Retention Status
Description: Percentage of participants with an adalimumab treatment status of continuous, early intermittent, late intermittent, permanently discontinued, or other. Continuous=initiated on adalimumab, had no treatment interruption period, still on treatment at study termination, and completed the study. Early intermittent=initiated on adalimumab 40 mg, treated every other week (EOW) for < 112 days (16 weeks) after initiation of treatment, with afterwards ≥ 1 treatment interruption period of ≥ 70 consecutive days, on treatment at study termination, and completed the study. Late intermittent=initiated on adalimumab 40 mg, treated EOW for ≥ 112 days (16 weeks) after initiation of treatment, with afterwards ≥ 1 treatment interruption period of at least 70 consecutive days, on treatment at study termination, and completed the study. Permanently discontinued=received ≥ 1 dose of adalimumab and stopped adalimumab treatment permanently. Other=participants not belonging to any of the previous groups.
Time Frame: Month 24/ Early Termination visit
Population: Intention to Treat (ITT) set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any follow-up data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 191
percentage of participants
  Continuous | 44.0
  Early intermittent | 2.6
  Late intermittent | 8.4
  Permanently discontinued | 38.7
  Other | 6.3

2. Secondary Outcome: Psoriasis Area and Severity Index (PASI): Mean Percentage Improvement From Baseline for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Four anatomic sites (head, upper extremities, trunk, and lower extremities) were assessed with PASI for erythema, induration (plaque thickness), and desquamation (scaling) as seen on the day of the examination. The severity of each sign was assessed using a 5-point scale: 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. PASI percentage improvement=100*(PASI score at Baseline - score at follow-up visit) / PASI score at Baseline. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: Baseline, TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730); last observation (up to 24 months)
Population: ITT set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any follow-up data were available; n=number of participants with an assessment at Baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage improvement
Groups:
- Participants Treated With Adalimumab: Continuous: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was 'continuous' (initiated on adalimumab, had no treatment interruption period, still on treatment at study termination, and completed the study).
- Participants Treated With Adalimumab: Early Intermittent: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was 'early intermittent' (initiated on adalimumab 40 mg, treated EOW for < 112 days [16 weeks] after initiation of treatment, with afterwards ≥ 1 treatment interruption period of ≥ 70 consecutive days, on treatment at study termination, and completed the study).
- Participants Treated With Adalimumab: Late Intermittent: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was 'late intermittent' (initiated on adalimumab 40 mg, treated EOW for ≥ 112 days [16 weeks] after initiation of treatment, with afterwards ≥ 1 treatment interruption period of at least 70 consecutive days, on treatment at study termination, and completed the study).
- Participants Treated With Adalimumab: Permanently Discontinued: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was 'permanently discontinued' (received ≥ 1 dose of adalimumab and stopped adalimumab treatment permanently).
- Participants Treated With Adalimumab: Other: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was 'other' (participants not belonging to any of the previous treatment status groups).
- Participants Treated With Adalimumab: All Participants: Participants with chronic plaque psoriasis in whom adalimumab (Humira) treatment was initiated and whose treatment status was one of the following: 'continuous,' early intermittent,' 'late intermittent,' 'permanently discontinued,' or 'other.'
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage improvement
  TW 3 months; n=76, 3, 16, 65, 9, 169 | 74.15 (27.06) | 95.69 (7.46) | 82.25 (13.78) | 49.96 (43.34) | 56.70 (24.05) | 65.06 (35.52)
  TW 12 months; n=69, 2, 13, 54, 8, 146 | 89.28 (13.73) | 33.00 (65.69) | 67.55 (26.79) | 52.35 (62.07) | 77.39 (12.15) | 72.26 (43.62)
  TW 24 months; n=77, 5, 15, 47, 3, 147 | 88.52 (17.06) | 42.46 (45.00) | 69.82 (28.62) | 75.93 (26.26) | 36.41 (58.03) | 79.96 (26.28)
  Last observation; n=80, 5, 16, 72, 11, 184 | 88.27 (17.06) | 42.46 (45.00) | 69.99 (27.66) | 67.63 (32.36) | 57.46 (38.94) | 75.52 (29.48)

3. Secondary Outcome: PASI: Percentage Improvement Change Categories From Baseline for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Percentage of participants who achieved ≥ 50%, 75%, 90% or 100% reduction (improvement) from Baseline in PASI score (PASI50, PASI75, PASI90, PASI100). Four anatomic sites (head, upper extremities, trunk, and lower extremities) were assessed for erythema, induration (plaque thickness), and desquamation (scaling) as seen on the day of the examination. The severity of each sign was assessed using a 5-point scale: 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. PASI percentage improvement=100*(PASI score at Baseline - score at follow-up visit) / PASI score at Baseline. For the purpose of analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based on the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: ITT set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any follow-up data were available; n=number of participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of participants
  TW 3 months: ≥ 50%; n=76, 3, 16, 65, 9, 169 | 85.5 | 100.0 | 100.0 | 64.6 | 55.6 | 77.5
  TW 3 months: ≥ 75%; n=76, 3, 16, 65, 9, 169 | 64.5 | 100.0 | 75.0 | 35.4 | 33.3 | 53.3
  TW 3 months: ≥ 90%; n=76, 3, 16, 65, 9, 169 | 26.3 | 66.7 | 31.3 | 15.4 | 0.0 | 21.9
  TW 3 months: = 100%; n=76, 3, 16, 65, 9, 169 | 5.3 | 66.7 | 12.5 | 7.7 | 0.0 | 7.7
  TW 12 months: ≥ 50%; n=69, 2, 13, 54, 8, 146 | 97.1 | 50.0 | 76.9 | 68.5 | 100.0 | 84.2
  TW 12 months: ≥ 75%; n=69, 2, 13, 54, 8, 146 | 85.5 | 50.0 | 30.8 | 40.7 | 62.5 | 62.3
  TW 12 months: ≥ 90%; n=69, 2, 13, 54, 8, 146 | 63.8 | 0.0 | 30.8 | 24.1 | 12.5 | 42.5
  TW 12 months: = 100%; n=69, 2, 13, 54, 8, 146 | 31.9 | 0.0 | 23.1 | 13.0 | 0.0 | 21.9
  TW 24 months: ≥ 50%; n=77, 5, 15, 47, 3, 147 | 94.8 | 60.0 | 73.3 | 87.2 | 66.7 | 88.4
  TW 24 months: ≥ 75%; n=77, 5, 15, 47, 3, 147 | 84.4 | 40.0 | 53.3 | 63.8 | 33.3 | 72.1
  TW 24 months: ≥ 90%; n=77, 5, 15, 47, 3, 147 | 66.2 | 0.0 | 33.3 | 34.0 | 0.0 | 49.0
  TW 24 months: = 100%; n=77, 5, 15, 47, 3, 147 | 39.0 | 0.0 | 13.3 | 8.5 | 0.0 | 24.5
  Last observation: ≥ 50%; n=80, 5, 16, 72, 11, 184 | 95.0 | 60.0 | 75.0 | 80.6 | 72.7 | 85.3
  Last observation: ≥ 75%; n=80, 5, 16, 72, 11, 184 | 83.8 | 40.0 | 50.0 | 52.8 | 45.5 | 65.2
  Last observation: ≥ 90%; n=80, 5, 16, 72, 11, 184 | 65.0 | 0.0 | 31.3 | 25.0 | 9.1 | 41.3
  Last observation: = 100%; n=80, 5, 16, 72, 11, 184 | 37.5 | 0.0 | 12.5 | 6.9 | 0.0 | 20.1

4. Secondary Outcome: Mean Percent Affected Body Surface Area (BSA) For All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Clinical psoriasis evaluations by the investigator of percentage of affected BSA. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of affected BSA
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of affected BSA
  Baseline; n=84, 5, 16, 71, 11, 187 | 21.92 (15.02) | 24.80 (23.19) | 18.25 (10.46) | 22.02 (15.54) | 23.95 (18.25) | 21.84 (15.21)
  Time-window 3 months; n=79, 3, 15, 66, 10, 173 | 7.67 (9.33) | 1.67 (2.89) | 4.34 (4.75) | 11.33 (13.57) | 15.16 (20.73) | 9.11 (11.89)
  Time-window 12 months; n=73, 1, 12, 54, 9, 149 | 2.83 (3.56) | 31.00 (NA) — Only 1 participant was assessed at this time point. | 2.25 (2.14) | 9.09 (13.44) | 4.44 (4.93) | 5.34 (9.27)
  Time-window 24 months; n=78, 5, 15, 45, 1, 144 | 1.71 (2.39) | 9.80 (6.61) | 4.88 (5.48) | 4.82 (6.73) | 1.00 (NA) — Only 1 participant was assessed at this time point. | 3.29 (5.01)
  Last Observation; n=84, 5, 16, 74, 12, 191 | 2.03 (3.06) | 9.80 (6.61) | 4.89 (5.29) | 6.42 (7.50) | 5.51 (5.27) | 4.39 (5.95)

5. Secondary Outcome: Physician's Global Assessment (PGA): Percentage of Participants in Regrouped PGA Categories for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: The PGA was an evaluation of a participant's psoriasis on a 6-point scale: clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5), which were then regrouped into the 2 categories "Clear/Minimal" or "Mild/Moderate/Severe/Very Severe (M/Md/S/VS)," and presented as the percentage of participants in each. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: Baseline, TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730); last observation (obs.; up to 24 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of participants
  Baseline: Clear/Minimal; n=82,5,16,73,12,188 | 1.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.5
  Baseline: M/Md/S/VS; n=82,5,16,73,12,188 | 98.8 | 100.0 | 100.0 | 100.0 | 100.0 | 99.5
  TW 3 months: Clear/Minimal; n=78,3,16,66,10,173 | 59.0 | 66.7 | 43.8 | 28.8 | 40.0 | 45.1
  TW 3 months: M/Md/S/VS; n=78,3,16,66,10,173 | 41.0 | 33.3 | 56.3 | 71.2 | 60.0 | 54.9
  TW 12 months: Clear/Minimal; n=73,1,12,54,9,149 | 78.1 | 0.0 | 33.3 | 35.2 | 22.2 | 55.0
  TW 12 months: M/Md/S/VS; n=73,1,12,54,9,149 | 21.9 | 100.0 | 66.7 | 64.8 | 77.8 | 45.0
  TW 24 months: Clear/Minimal; n=81,5,15,47,1,149 | 77.8 | 0.0 | 46.7 | 36.2 | 0.0 | 58.4
  TW 24 months: M/Md/S/VS; n=81,5,15,47,1,149 | 22.2 | 100.0 | 53.3 | 63.8 | 100.0 | 41.6
  Last obs.: Clear/Minimal; n=84,5,16,74,12,191 | 77.4 | 0.0 | 43.8 | 32.4 | 16.7 | 51.3
  Last obs.: M/Md/S/VS; n=84,5,16,74,12,191 | 22.6 | 100.0 | 56.3 | 67.6 | 83.3 | 48.7

6. Secondary Outcome: Dermatology Life Quality Index (DLQI): Mean Score for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: DLQI score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each question are: very much (3), a lot (2), a little (1), or not at all (0). The total DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows, based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
units on a scale
  Baseline; n=80, 5, 15, 70, 12, 182 | 12.48 (7.18) | 13.80 (6.72) | 12.27 (6.13) | 12.97 (7.02) | 12.08 (7.35) | 12.66 (6.97)
  Time-window 3 months; n=73, 3, 15, 61, 8, 160 | 3.41 (4.69) | 0.33 (0.58) | 3.53 (5.80) | 5.38 (5.89) | 7.13 (9.51) | 4.30 (5.62)
  Time-window 12 months; n=68, 1, 12, 47, 6, 134 | 1.51 (2.33) | 18.00 (NA) — Only 1 participant was assessed at this time point. | 3.42 (3.03) | 6.94 (6.54) | 3.33 (6.31) | 3.79 (5.24)
  Time-window 24 months; n=71, 5, 14, 44, 3, 137 | 1.44 (3.21) | 7.40 (3.51) | 5.50 (5.17) | 4.32 (5.42) | 10.00 (9.00) | 3.18 (4.79)
  Last Observation; n=82, 5, 15, 74, 12, 188 | 1.56 (3.19) | 7.40 (3.51) | 5.13 (5.18) | 6.08 (6.74) | 8.25 (8.40) | 4.21 (5.87)

7. Secondary Outcome: DLQI: Percentage of Participants in DLQI Categories for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: DLQI is a participant-reported outcome consisting of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot (score of 2), a little (score of 1), or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. The following scoring categories present the effect on participant's life: 0-1 no effect at all; 2-5 small effect; 6-10 moderate effect; 11-20 very large effect; 21-30 extremely large effect. Follow-up visits were classified into time windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of participants
  Baseline: score 0-1; n=80,5,15,70,12,182 | 5.0 | 0.0 | 6.7 | 2.9 | 16.7 | 4.9
  Baseline: score 2-5; n=80,5,15,70,12,182 | 12.5 | 0.0 | 6.7 | 15.7 | 0.0 | 12.1
  Baseline: score 6-10; n=80,5,15,70,12,182 | 27.5 | 40.0 | 20.0 | 15.7 | 25.0 | 22.5
  Baseline: score 11-20; n=80,5,15,70,12,182 | 41.3 | 40.0 | 46.7 | 51.4 | 50.0 | 46.2
  Baseline: score 21-30; n=80,5,15,70,12,182 | 13.8 | 20.0 | 20.0 | 14.3 | 8.3 | 14.3
  TW 3 months: score 0-1; n=73,3,15,61,8,160 | 50.7 | 100.0 | 46.7 | 27.9 | 50.0 | 42.5
  TW 3 months: score 2-5; n=73,3,15,61,8,160 | 26.0 | 0.0 | 33.3 | 34.4 | 12.5 | 28.8
  TW 3 months: score 6-10; n=73,3,15,61,8,160 | 16.4 | 0.0 | 6.7 | 19.7 | 12.5 | 16.3
  TW 3 months: score 11-20; n=73,3,15,61,8,160 | 5.5 | 0.0 | 6.7 | 16.4 | 12.5 | 10.0
  TW 3 months: score 21-30; n=73,3,15,61,8,160 | 1.4 | 0.0 | 6.7 | 1.6 | 12.5 | 2.5
  TW 12 months: score 0-1; n=68,1,12,47,6,134 | 69.1 | 0.0 | 41.7 | 31.9 | 66.7 | 53.0
  TW 12 months: score 2-5; n=68,1,12,47,6,134 | 26.5 | 0.0 | 33.3 | 17.0 | 16.7 | 23.1
  TW 12 months: score 6-10; n=68,1,12,47,6,134 | 2.9 | 0.0 | 25.0 | 19.1 | 0.0 | 10.4
  TW 12 months: score 11-20; n=68,1,12,47,6,134 | 1.5 | 100.0 | 0.0 | 27.7 | 16.7 | 11.9
  TW 12 months: score 21-30; n=68,1,12,47,6,134 | 0.0 | 0.0 | 0.0 | 4.3 | 0.0 | 1.5
  TW 24 months: score 0-1; n=71,5,14,44,3,137 | 76.1 | 0.0 | 35.7 | 47.7 | 33.3 | 59.1
  TW 24 months: score 2-5; n=71,5,14,44,3,137 | 16.9 | 40.0 | 21.4 | 15.9 | 0.0 | 17.5
  TW 24 months: score 6-10; n=71,5,14,44,3,137 | 4.2 | 40.0 | 21.4 | 27.3 | 33.3 | 15.3
  TW 24 months: score 11-20; n=71,5,14,44,3,137 | 2.8 | 20.0 | 21.4 | 6.8 | 33.3 | 7.3
  TW 24 months: score 21-30; n=71,5,14,44,3,137 | 0.0 | 0.0 | 0.0 | 2.3 | 0.0 | 0.7
  Last observation: score 0-1; n=82,5,15,74,12,188 | 73.2 | 0.0 | 40.0 | 37.8 | 41.7 | 52.7
  Last observation: score 2-5; n=82,5,15,74,12,188 | 18.3 | 40.0 | 20.0 | 14.9 | 0.0 | 16.5
  Last observation: score 6-10; n=82,5,15,74,12,188 | 6.1 | 40.0 | 20.0 | 27.0 | 25.0 | 17.6
  Last observation: score 11-20; n=82,5,15,74,12,188 | 2.4 | 20.0 | 20.0 | 16.2 | 25.0 | 11.2
  Last observation: score 21-30; n=82,5,15,74,12,188 | 0.0 | 0.0 | 0.0 | 4.1 | 8.3 | 2.1

8. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire: Mean Percentage of Work Time Missed (Absenteeism) for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Absenteeism, presented as the mean percentage of work time missed due to psoriasis (as reported on the WPAI), and calculated as: 100*number of hours of work missed due to psoriasis / (number of hours of work missed due to psoriasis + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: ITT set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any follow-up data were available; n=number of participants with assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of work time missed
  Baseline; n=48, 4, 9, 35, 10, 106 | 3.05 (14.92) | 25.00 (50.00) | 0.00 (0.00) | 2.92 (16.90) | 1.00 (2.27) | 3.38 (16.83)
  Time-window 3 months; n=43, 2, 7, 31, 6, 89 | 0.21 (1.39) | 0.00 (0.00) | 0.00 (0.00) | 0.81 (4.49) | 0.86 (2.11) | 0.44 (2.85)
  Time-window 12 months; n=39, 1, 5, 26, 3, 74 | 0.00 (0.00) | 0.00 (NA) — Only 1 participant had an assessment at this time point. | 0.00 (0.00) | 0.00 (0.00) | 17.78 (30.79) | 0.72 (6.20)
  Time-window 24 months; n=41, 4, 11, 22, 0, 78 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 2.27 (10.66) | NA (NA) — No participants had an assessment at this time point. | 0.64 (5.66)
  Last observation; n=60, 4, 11, 47, 11, 133 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 2.66 (10.73) | 6.62 (16.10) | 1.49 (7.98)

9. Secondary Outcome: WPAI Questionnaire: Mean Percentage of Impairment While Working Due to Psoriasis (Presenteeism) for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Presenteeism (the extent to which psoriasis decreased productivity) is presented as the mean percentage of impairment while working due to psoriasis, and calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: ITT set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any follow-up data were available.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of impairment while working
  Baseline; n=52, 3, 9, 37, 10, 111 | 22.50 (25.81) | 0.00 (0.00) | 11.11 (11.67) | 18.51 (19.82) | 30.00 (19.44) | 20.32 (22.55)
  Time-window 3 months; n=46, 2, 8, 34, 6, 96 | 6.74 (18.26) | 0.00 (0.00) | 0.00 (0.00) | 6.18 (13.71) | 28.33 (38.17) | 7.19 (18.28)
  Time-window 12 months; n=45, 1, 6, 27, 3, 82 | 4.22 (12.34) | 60.00 (NA) — Only 1 participant had an assessment at this time point. | 5.00 (8.37) | 9.26 (17.30) | 10.00 (17.32) | 6.83 (15.22)
  Time-window 24 months; n=46, 4, 11, 24, 0, 85 | 2.61 (8.01) | 12.50 (25.00) | 16.36 (21.57) | 5.42 (10.21) | NA (NA) — No participants had an assessment at this time point. | 5.65 (12.77)
  Last observation; n=60, 4, 11, 49, 11, 135 | 3.33 (8.77) | 12.50 (25.00) | 16.36 (21.57) | 9.08 (19.03) | 20.91 (27.37) | 8.19 (17.27)

10. Secondary Outcome: WPAI Questionnaire: Mean Percentage of Total Work Productivity Impairment (TWPI) Due to Psoriasis for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: The mean percentage of TWPI due to psoriasis (based on the WPAI questionnaire) is presented, calculated as: Absenteeism (%) + extent to which psoriasis decreased productivity (%)* [number of hours worked / (number of hours of work missed due to psoriasis + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: ITT set: all participants enrolled in the study who received at least 1 dose of adalimumab, and for whom any data follow-up were available; n=number of participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of TWPI
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of TWPI
  Baseline; n=47, 3, 9, 34, 10, 103 | 21.29 (25.24) | 0.00 (0.00) | 11.11 (11.67) | 16.78 (16.71) | 30.64 (19.42) | 19.20 (21.33)
  Time-window 3 months; n=42, 2, 7, 31, 6, 88 | 6.65 (18.82) | 0.00 (0.00) | 0.00 (0.00) | 6.69 (15.40) | 28.42 (38.33) | 7.47 (19.23)
  Time-window 12 months; n=39, 1, 5, 26, 3, 74 | 3.85 (11.84) | 60.00 (NA) — 1 participant had an assessment at this time point. | 2.00 (4.47) | 9.62 (17.55) | 27.78 (26.74) | 7.48 (16.26)
  Time-window 24 months; n=41, 4, 11, 22, 0, 78 | 2.20 (7.25) | 12.50 (25.00) | 16.36 (21.57) | 7.27 (13.86) | NA (NA) — No participants had an assessment at this time point. | 6.15 (13.79)
  Last observation; n=60, 4, 11, 47, 11, 133 | 3.83 (10.10) | 12.50 (25.00) | 16.36 (21.57) | 9.95 (19.14) | 26.58 (28.68) | 9.17 (18.11)

11. Secondary Outcome: WPAI Questionnaire: Mean Percentage of Activity Impairment Due to Psoriasis for All Participants and Broken Down by Adalimumab Treatment Retention Status
Description: Activity impairment due to psoriasis (the extent to which psoriasis affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. For the purpose of the analysis of the evolution of parameters over time, follow-up visits were classified into time-windows (TWs), based upon the number of days between onset of adalimumab treatment and the date of each subsequent visit: TW 3 months=period between Day 1 and 137 (target, Day 91); TW 12 months=period between Day 275 and 456 (target, Day 365); TW 24 months=period starting on Day 640 (target Day 730).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Participants Treated With Adalimumab: Continuous | Participants Treated With Adalimumab: Early Intermittent | Participants Treated With Adalimumab: Late Intermittent | Participants Treated With Adalimumab: Permanently Discontinued | Participants Treated With Adalimumab: Other | Participants Treated With Adalimumab: All Participants
Number analyzed (Participants) | 84 | 5 | 16 | 74 | 12 | 191
percentage of activity impairment
  Baseline; n=74, 5, 13, 65, 10, 167 | 33.38 (28.05) | 28.00 (31.14) | 32.31 (23.86) | 34.92 (26.35) | 35.00 (20.68) | 33.83 (26.52)
  Time-window 3 months; n=61, 3, 13, 57, 7, 141 | 8.36 (16.35) | 0.00 (0.00) | 8.46 (14.05) | 20.53 (28.37) | 40.00 (41.63) | 14.68 (24.48)
  Time-window 12 months; n=63, 1, 11, 43, 5, 123 | 5.56 (13.65) | 40.00 (NA) — Only 1 participant had an assessment at this time point. | 12.73 (16.18) | 17.91 (24.35) | 10.00 (14.14) | 10.98 (19.14)
  Time-window 24 months; n=64, 5, 14, 40, 2, 125 | 4.53 (13.68) | 32.00 (39.62) | 18.57 (19.94) | 12.00 (18.43) | 25.00 (35.36) | 9.92 (18.77)
  Last observation; n=82, 5, 15, 73, 10, 185 | 4.02 (12.26) | 32.00 (39.62) | 17.33 (19.81) | 17.40 (25.61) | 21.00 (29.98) | 12.05 (22.09)

ADVERSE EVENTS:
Time Frame: From informed consent through Month 24 (or early termination) + 70 days after the date of last administration of adalimumab. Mean (SD) study duration: 23.18 (5.64) months.
Arm/Group | Participants Treated With Adalimumab
Serious Adverse Events (participants affected / at risk) | 19/191
Other Adverse Events (participants affected / at risk) | 67/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Treated With Adalimumab (N=191)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Aplasia (Congenital, familial and genetic disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Ocular icterus (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Drug ineffective (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 2
Malaise (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Immunodeficiency (Immune system disorders) | 1
Lung infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Double stranded DNA antibody positive (Investigations) | 1
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back disorder (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Activities of daily living impaired (Social circumstances) | 1
Treatment noncompliance (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Treated With Adalimumab (N=191)
Drug ineffective (General disorders) | 36
Injection site pain (General disorders) | 2
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 2
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.